CLINICAL TRIAL: NCT00750516
Title: Lactic Acid Levels In Hypotensive Patients Without(Standard) and With Tourniquet
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient patient enrolled
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Susan Wojcik, Associate Professor, State University of New York - Upstate Medical University
Other Study IDs: 5625
Record Dates: First submitted 2008-09-09; First posted 2008-09-10 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Hypotension; Sepsis
Keywords: Lactic acid; hypotension; sepsis
MeSH Terms: conditions — Hypotension; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lacid: Hypotensive, non pregnant by history, non comfort care Emergency Department patients.

SUMMARY:
This study seeks to determine whether the Lactic Acid blood level in a critically ill patient must be drawn with a non-tourniquet venipuncture. The null hypothesis is that there is no significant difference in Lactic Acid blood level in critically ill patients in a sample taken from either with a tourniquet or a non-tourniquet veni-puncture.

Monitoring of Lactic acid level is helpful in both identifying potentially serious ill patients as well as identifying in the ICU patients with high morbidity and mortality.

When a patient arrives to an Emergency Department and that patient is hypotensive (BP less than or equal to 90 systolic), the nursing staff often starts an IV and if possible draws the patient's initial blood tests off that first IV site; or if the patient has had an IV started in the field by EMS, the nursing staff will draw blood from another site using a tourniquet. This initial work up by the nursing staff takes 15 -20 minutes before a physician may see the patient. Since the present standard Lactic Acid test must be drawn either by arterial puncture or venipuncture without a tourniquet, this test is rarely done as part of their (the RNs) initial blood draws.

This simple impediment of needing to repeat the venipuncture without a tourniquet, especially in patients who often have venous access difficulty, delays the identification of appropriate patients for early and aggressive management- particularly those with sepsis.

Our hypothesis is that this requirement for a non-tourniquet blood draw is unnecessary.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure systolic of 90 or less
* Non pregnant by history

Exclusion Criteria:

* Pregnant by history
* Comfort care only

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypotensive, non pregnant by history, Emergency Medicine patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Differences in hypotensive patients between the use of a tourniquet and non tourniquet sampling for Lactic Acid level. | At the initial evaluation of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Mark Barasz, MD, Principal Investigator — Emergency Medicine Department ofUpstate Hospital
Locations (1):
- Upstate Hospital Emergency Department, Syracuse, New York, United States